CLINICAL TRIAL: NCT00289887
Title: A Double-Blind, Randomized, Parallel, Efficacy Study Evaluating Losartan Potassium Alone or in Combination With Hydrochlorothiazide Versus Placebo in Obese Patients With Elevated Systolic and Diastolic Blood Pressure
Brief Title: Obese Hypertension Study (0954-315)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0954-315; MK0954-315; 2006_002
Record Dates: First submitted 2006-02-08; First posted 2006-02-10 (Estimated); Results first posted 2010-05-27 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Losartan
  Interventions: Drug: Comparator: losartan +/- HCTZ
- 2 (Placebo Comparator): Placebo
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: Comparator: losartan +/- HCTZ — Placebo to losartan once daily for 4 weeks in run-in period. Then, losartan 50 mg for 4 weeks, then titrate to losartan 100 mg at Week 4, then titrate to losartan 100 mg + hydrochlorothiazide (HCTZ) 12.5 mg at Week 8, and finally titrate to losartan 100 mg + HCTZ 25 mg at Week 12. Duration of treatment is approximately 16 weeks.
  Arms: 1
Drug: Comparator: Placebo — Placebo to losartan once daily for 4 weeks in run-in period. Then, placebo to losartan or losartan/HCTZ once daily for approximately 16 weeks.
  Arms: 2

SUMMARY:
This is a 16-week study to evaluate high systolic and diastolic blood pressure following treatment in obese, hypertensive, adult patients.

ELIGIBILITY:
Inclusion Criteria:

* Obese male and female patients, ages 21-75 years, with high blood pressure

Exclusion Criteria:

* Patients cannot have any other severe cardiac conditions

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 261 (Actual)
Dates: Start 2006-02; Primary Completion 2007-02 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Oparil S, Abate N, Chen E, Creager MA, Galet V, Jia G, Julius S, Lerman A, Lyle PA, Pool J, Tershakovec AM. A double-blind, randomized study evaluating losartan potassium monotherapy or in combination with hydrochlorothiazide versus placebo in obese patients with hypertension. Curr Med Res Opin. 2008 Apr;24(4):1101-14. doi: 10.1185/030079908x280716. Epub 2008 Mar 6. PMID 18328120

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited at 51 sites in the United States.
  Prime Therapy Period: April 2006 to February 2007
Pre-assignment Details: Prior antihypertensive medications were withdrawn/ tapered before patients entered the 4-week placebo run-in period.
Groups:
- Losartan: Once-daily losartan 50 mg titrated at 4-week intervals to losartan 100 mg, losartan 100 mg/Hydrochlorothiazide (HCTZ) 12.5 mg, and losartan 100 mg/HCTZ 25 mg
- Placebo: Once-daily matching placebo for losartan 50 mg titrated at 4-week intervals to matching placebo for losartan 100 mg, matching placebo for losartan 100 mg/HCTZ 12.5 mg, and matching placebo for losartan 100 mg/HCTZ 25 mg
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 127 | 134
Completed | 105 | 105
Not Completed | 22 | 29
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 3 | 11
Not completed — Lost to Follow-up | 3 | 3
Not completed — Protocol Violation | 3 | 1
Not completed — Withdrawal by Subject | 3 | 8
Not completed — Other | 7 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 127 | 134 | 261
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.1 (10.4) | 51.4 (9.7) | 50.8 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 77 | 156
  Male | 48 | 57 | 105
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 84 | 87 | 171
  Black | 22 | 29 | 51
  Hispanic American | 20 | 16 | 36
  Native American | 0 | 1 | 1
  Other | 1 | 1 | 2
Sitting Diastolic Blood Pressure (SiDBP) [Mean (Standard Deviation); unit: mm Hg] | 99.1 (4.2) | 99.0 (4.0) | 99.0 (4.1)
Sitting Systolic Blood Pressure (SiSBP) [Mean (Standard Deviation); unit: mm Hg] | 151.6 (8.2) | 152.4 (9.0) | 152.0 (8.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) at Week 8
Description: Mean change from baseline in trough (6 hours after last morning dose) SiSBP at Week 8.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 8 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: An "all patients treated" approach was employed, patients included had at least 1 dose post baseline and 1 measurement at baseline and during treatment.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 119 | 117
mm Hg | -12.1 (1.2) | -6.8 (1.2)

2. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 8
Description: Mean change from baseline in trough (6 hours after the last morning dose) SiDBP at Week 8.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 8 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 119 | 117
mm Hg | -9.7 (0.8) | -6.9 (0.8)

3. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 12
Description: Mean change from baseline in trough (6 hours after the last morning dose) SiDBP at Week 12.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 12 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 109 | 112
mm Hg | -12.9 (0.8) | -7.1 (0.8)

4. Primary Outcome: Mean Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) at Week 12
Description: Mean change from baseline in trough (6 hours after last morning dose) SiSBP at Week 12.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 12 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 109 | 112
mm Hg | -16.7 (1.3) | -6.8 (1.3)

5. Primary Outcome: Mean Change From Baseline in Trough Sitting Systolic Blood Pressure (SiSBP) at Week 16
Description: Mean change from baseline in trough (6 hours after last morning dose) SiSBP at Week 16.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 16 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 106 | 106
mm Hg | -19.1 (1.3) | -6.4 (1.3)

6. Primary Outcome: Mean Change From Baseline in Trough Sitting Diastolic Blood Pressure (SiDBP) at Week 16
Description: Mean change from baseline in trough (6 hours after the last morning dose) SiDBP at Week 16.
  A mixed effects model (with repeated measurements including terms of treatment, investigators, week, baseline SiSBP(/SiDBP), plasma glucose stratum, treatment*week, and week*SiSBP(/SiDBP)) was used to compare the treatments on the change from baseline.
Time Frame: At baseline and at 16 weeks (with the measurements taken prior to the morning dose, between 6 AM and 10 AM)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 106 | 106
mm Hg | -14.1 (0.9) | -6.0 (0.9)

ADVERSE EVENTS:
Time Frame: Week 0 through Week 16.
Arm/Group | Losartan | Placebo
Serious Adverse Events (participants affected / at risk) | 1/127 | 1/134
Other Adverse Events (participants affected / at risk) | 4/127 | 7/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan (N=127) | Placebo (N=134)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Losartan (N=127) | Placebo (N=134)
Headache (Nervous system disorders) | 4 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.